CLINICAL TRIAL: NCT00254280
Title: Treatment of Recalcitrant Hand and Foot Warts With Intense Pulsed Light and Paring Versus Paring Alone - a Randomized Controlled Trial With Blinded Response Evaluation
Brief Title: Treatment of Recalcitrant Hand and Foot Warts With Intense Pulsed Light - a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KF-01-255566
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Warts
Keywords: Warts; Intense pulsed light; RCT; Recalcitrant hand and foot warts
MeSH Terms: conditions — Warts

INTERVENTIONS:
Procedure: Intense Pulsed Light + paring versus paring alone

SUMMARY:
The purpose of the study is for recalcitrant hand and foot warts to compare the efficacy of treatment with Intense Pulsed Light and paring versus paring alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Recalcitrant warts
* No previous IPL treatment of warts

Exclusion Criteria:

* Immunosuppressive treatment
* Patients suffering from HIV, diabetes or other immunosuppressive diseases
* Pregnancy
* Previous IPL treatment
* Patients with a tendency to prodyce keloids or hypertrophic scars
* Mosaic and flat warts
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-11; Study Completion 2008-09

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, PhD, DrMedSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg hospital, Copenhagen, Copenhagen NV, Denmark